CLINICAL TRIAL: NCT03091010
Title: A Comparison of Fecal Microbiota Transplantation and Steroid Therapy in Patients With Severe Alcoholic Hepatitis A Randomized Controlled Trial.
Brief Title: A Comparison of Fecal Microbiota Transplantation and Steroid Therapy in Patients With Severe Alcoholic Hepatitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Alcoholic Hepatitis-01
Record Dates: First submitted 2017-03-09; First posted 2017-03-27 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-10

CONDITIONS: Severe Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Fecal Microbiota Transplantation; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplantation (Experimental)
  Interventions: Other: Fecal Microbiota Transplantation
- Steroid (Active Comparator)
  Interventions: Drug: Steroids

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation will be given 100mL of suspension. It will given for a period of 7 days
  Arms: Fecal Microbiota Transplantation
Drug: Steroids — Oral steroids 40 mg (prednisolone) will be given for a period of 7 days in hospital followed by 3 weeks on OPD basis
  Arms: Steroid

SUMMARY:
Study population: Patients attending the Out Patient Department and admitted to Institute of Liver and Biliary Sciences.

Study design: Prospective randomized controlled trial Study period: One year- January 2017- December 2018 Sample size: 130 (65 cases in each group) Intervention: The subjects will be given Fecal Microbiota Transplantation through a NJ tube placed after admission to the hospital. Participants will be administered the processed fecal microbiota sample collected from a related or unrelated healthy donor for a period of 7 days.

Monitoring and assessment:

The recipient will be monitored every day after Fecal Microbiota Transplantation therapy.

The recipient will undergo physical examination, complete blood counts, at baseline and a chest X ray, serum procalcitonin, CRP and Tumor Necrosis Factor alpha levels, Liver Function Tests, Kidney Function Tests, International Normalized Ratio and arterial ammonia, at day 0,4,7,14,28,90,180,270 and 365 from the start of therapy.

Microbiota analysis of the donors will be done at baseline and the recipients will be done on day 0,7,28,90 & 180.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe alcoholic hepatitis .
* Eligible for steroid therapy.

Exclusion Criteria:

* Upper gastrointestinal bleed within the past one month.
* Active sepsis
* Serum creatinine > 1.5 mg/dl (Hepato renal syndrome)
* Intestinal paralysis
* Hepatic or extrahepatic malignancy
* Disseminated intravascular coagulation
* Discriminant Function (DF) >90

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-04-08 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Overall Survival at 3 months | 3 months

SECONDARY OUTCOMES:
Improvement in Child Pugh Turcotte (score) severity in both groups | 6 months
Improvement in Model for End Stage Liver Disease (MELD) of liver disease severity in both groups | 6 months
Improvement in Glasgow Alcoholic Hepatitis (score) in both groups | 6 months
Improvement in Maddrey's Discriminant Function (score) in both groups | 6 months
Adverse events in both groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No